CLINICAL TRIAL: NCT00480064
Title: Randomized Prospective Study of Adding Lomustine to Idarubicin and Cytarabine for Induction Chemotherapy and Adding Intermediate Dose Cytarabine to Consolidation in Older Patients With Acute Myeloid Leukaemia
Brief Title: Lomustine and Intermediate Dose Cytarabine in Older Patients With AML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGMT95-V
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; older patients; lomustine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lomustine, intermediate dose cytarabine

SUMMARY:
A multicenter randomized trial was performed comparing induction therapy (IC: Idarubicin and Cytarabine, 5+7) to ICL (the same drugs plus lomustine (CCNU), 200mg\m2 orally at day 1). Patients in complete remission (CR) were then randomized to receive either maintenance therapy or intensification with intermediate-dose cytarabine and idarubicin followed by maintenance therapy.

DETAILED DESCRIPTION:
Induction therapy: Patients were randomized to receive idarubicin plus cytarabine (IC) or the same drugs plus lomustine (ICL), the latter given at the dose of 200 mg/m2 orally at day 1. Patients with persistent leukemia in the bone marrow, defined by at least 20% marrow cellularity with more than 5% blasts on day 14 or at a subsequent time point following initiation of induction therapy, received a second course of induction chemotherapy identical to the initial induction course. Non-responders to the second induction course were taken off the protocol.

Consolidation therapy: After completing induction treatment, patients who were in complete remission after 1 or 2 induction courses received a course of consolidation (IC') therapy with idarubicin and subcutaneous cytarabine. Subsequently, if stable remission persisted, the patients received maintenance therapy or maintenance therapy preceded by a second consolidation (IIC) with intermediate-dose cytarabine. Randomization was performed as soon as CR was achieved.

Maintenance therapy: This was conducted in all patients with persisting CR one month after completing the first (IC) or second (IIC) consolidation and consisted of the following: five courses of combination chemotherapy at 1, 3, 6, 9 and 13 months from the last consolidation, namely cytarabine (subcutaneously) and idarubicin and between these courses for one year: a continuous regimen of methotrexate and 6-mercaptopurine, as alternating 10 day-courses .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 years and older with de novo AML according to FAB criteria
* With normal cardiac function with left ventricular ejection fraction >= 50%, absence of unstable cardiac arrhythmia or unstable angina.
* Unimpaired renal (creatinin <180µmol\L)
* Unimpaired liver (bilirubin <35µmol\L) functions.
* Performance status <3
* Signed and dated informed consent.

Exclusion Criteria:

* Acute promyelocytic leukemia
* Patients with myeloproliferative syndromes prior to diagnosis of AML
* Patients who previously had myelodysplastic syndrome
* Patients pretreated with chemo- or radiotherapy
* Performance status <2
* Positive serology for HIV

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 1995-07; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Primary Outcomes: The primary objective of this study was to assess the ability of lomustine to increase the CR rate and to improve overall survival | 13 months

SECONDARY OUTCOMES:
Secondary Outcomes: The secondary objective was to test intermediate-dose cytarabine on survival, and to analyze the impact of prognostic factors on CR and survival. | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: JOSY REIFFERS, MD, Principal Investigator — CHU Haut-Leveque Pessac 33604 France
Locations (1):
- Josy REIFFERS, MD MS, Pessac, France